CLINICAL TRIAL: NCT01408615
Title: Post Marketing Surveillance for General Drug Use to Assess the Safety and Efficacy Profile of ELONVA in Usual Practice
Brief Title: A Post Marketing Observational Study of the Safety and Efficacy of Elonva (Corifollitropin Alfa) in General Practice (P08165)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P08165
Record Dates: First submitted 2011-06-02; First posted 2011-08-03 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: Women undergoing COS in combination with a GnRH antagonist for the development of multiple follicles in an ART program.
  Interventions: Drug: corifollitropin alfa

INTERVENTIONS:
Drug: corifollitropin alfa — 100 or 150 microgram single subcutaneous injection
  Other Names: Elonva

SUMMARY:
This observational study will examine the safety and efficacy profile of Elonva (corifollitropin alfa) when administered in Korean women undergoing controlled ovarian stimulation (COS) in combination with a gonadotropin-releasing hormone (GnRH) antagonist for the development of multiple follicles in an assisted reproductive technology (ART) program.

ELIGIBILITY:
Inclusion Criteria:

- Women with an indication for COS prior to in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) who meet the criteria as mentioned in the current Korean ELONVA local label

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Tumors of the ovary, breast, uterus, pituitary or hypothalamus
* Abnormal (not menstrual) vaginal bleeding without a known/diagnosed cause.
* Primary ovarian failure
* Ovarian cysts or enlarged ovaries
* A history of OHSS
* A previous COS cycle that resulted in more than 30 follicles ≥ 11 mm measured by ultrasound examination
* Basal antral follicle count > 20
* Fibroid tumors of the uterus incompatible with pregnancy
* Malformations of the reproductive organs incompatible with pregnancy
* Pregnancy
* Polycystic ovarian syndrome

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women participating in an ART program consisting of COS in combination with a GnRH antagonist in a general clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Oocytes Retrieved | At time of oocyte retrieval (up 3 days from human chorionic gonadotropin [hCG] injection)
Number of Participants who Experience Ovarian Hyperstimulation Syndrome (OHSS) | During treatment and up to 30 days after cessation of treatment
Number of Participants who report an serious adverse event (SAE) | During treatment and up to 30 days after cessation of treatment
Number of Participants who report an adverse event (AE) | During treatment and up to 30 days after cessation of treatment